CLINICAL TRIAL: NCT02412540
Title: A Parallel Cohort Controlled Trial of Outcome of Nonalcoholic Steatohepatitis in Adolescents After Bariatric Surgery vs. Comprehensive Lifestyle Intervention (NASH ABC)
Brief Title: Controlled Trial of WLS vs. CLI for Severely Obese Adolescents With NASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NASH ABC
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight Loss Surgery (No Intervention): Adolescents who will have Weight Loss Surgery and had biopsy-confirmed NASH. The Weight Loss Surgery is not part of the study. The investigators are following the adolescents after the surgery.
- Comprehensive Lifestyle Intervention (Experimental): Comprehensive Lifestyle Intervention - Dietary, activity and behavioral interventions. Adolescents who have biopsy-confirmed NASH and wish to participate in a Comprehensive Lifestyle Intervention (26+ contact hours) including individual meetings with a study dietitian, group nutrition classes, behavior management modules and physical activity goals.
  Interventions: Behavioral: Comprehensive Lifestyle Intervention

INTERVENTIONS:
Behavioral: Comprehensive Lifestyle Intervention — Dietary, behavioral and activity interventions designed to reduce weight.
  Arms: Comprehensive Lifestyle Intervention

SUMMARY:
The goal of this study is to determine effective treatment and identify diagnostic biomarkers for Nonalcoholic steatohepatitis (NASH). Individuals that take part in the study will be participating in either a weight loss surgery (WLS) group or a comprehensive lifestyle intervention (CLI) group. People in the WLS group will receive vertical sleeve gastrectomy (VSG). The CLI group will receive dietary, activity and behavioral interventions provided by trained study staff.

DETAILED DESCRIPTION:
The investigators have designed a rigorously controlled study designed to evaluate NASH outcomes in two parallel cohorts: 1) severely obese adolescents with NASH who have chosen to undergo WLS (specifically VSG) for clinical indications compared to 2) a control group of severely obese adolescents with NASH enrolled in a CLI offered as part of this study. The study will provide the best evidence to date of the effectiveness of WLS and CLI in treating NASH in adolescents with body mass index (BMI) ≥ 35 kg/m2. The investigators will also concurrently collect health-care utilization data to enable subsequent cost-effectiveness analyses (CEA) to evaluate the cost-effectiveness of WLS vs. CLI intervention in severely-obese adolescents with NASH. If the investigators' data support our hypothesis that WLS yields superior results, this will set the stage for randomized studies (if needed) and translational studies of weight loss-independent biological mechanism(s) unique to WLS, which may include specific changes in bile acid signaling and in the intestinal microbiome. The latter would facilitate developing novel pharmacotherapies accessible to younger or less obese children with NASH to whom WLS is not applicable. Cumulatively, this study has the potential to yield significant improvements in medical and quality of life (QOL) outcomes for a large proportion of pediatric patients with NASH and to reduce long term health care costs by identifying effective treatment options and decreasing progression to cirrhosis and end-stage liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 12-19 years (range as defined by World Health Organization).
* BMI ≥ 35 to 69 kg/m2 (minimum BMI per current guidelines for WLS in adolescents). An upper limit of BMI was set to avoid rare outliers in BMI.
* Meet current standard of care eligibility criteria for adolescent WLS.
* Liver biopsy for clinical indication to evaluate for NASH within 1 year of enrollment. Biopsy must confirm definite or borderline NASH with a minimum histological NASH Activity Score of ≥ 3.
* No evidence of any other liver disease by history, screening tests or histological evaluation.
* Written informed consent from parent/legal guardian and informed assent from the adolescent

Exclusion Criteria:

* Evidence of other chronic liver disease: autoimmune hepatitis; hepatitis B; hepatitis C; hemochromatosis; alpha-1-antitrypsin (A1AT) deficiency; Wilson disease; use of medications known to cause fatty liver for > 2 consecutive weeks in past year (i.e. systemic glucocorticoids, tetracycline, anabolic steroids, valproic acid); alcohol intake >10 gm/day females & >20 gm/day males.
* Non-compensated liver disease with any of the following: hemoglobin <10 g/dL; white blood cell count <3,500 cells/mm3, platelet count <130,000 cells/mm3 of blood, direct bilirubin >1.0 mg/dL, total bilirubin >3 mg/dL, albumin <3.2 g/dL, international normalized ratio (INR) >1.4
* Active psychiatric disorder that would prevent eligibility for WLS or impede adherence to CLI, including clinically significant depression (hospitalization or suicidal ideation) in past 12 months.
* Any medical condition preventing eligibility for WLS including but not limited to micronutrient deficiencies (e.g. iron) refractory to medical therapy or inflammatory bowel disease.
* Poorly controlled Type 2 diabetes mellitus (T2DM) defined as hemoglobin A1C (HgbA1c) > 10%.
* Initiation of high dose vitamin E (>400 IU per day) or other medications which could alter NASH histology at any time after baseline liver biopsy or during the trial. Stable dose of vitamin E that was started 12 months or more prior to biopsy is allowed.
* Weight reduction of >5% between baseline liver biopsy and enrollment, as weight loss >5% may change NASH severity.
* Inability or failure to provide informed assent/consent
* Current enrollment in another clinical trial or receipt of an investigational study drug within 6 months prior to the baseline liver biopsy
* Any female who is currently nursing, planning a pregnancy, known or suspected to be pregnant, or has a positive pregnancy screen
* Inability to travel to study site at intervals necessary for clinical interventions (CLI or WLS).
* Prior history of WLS.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Histology Endpoint: Proportion of subjects achieving greater than 2 point reduction in NASH activity score (NAS) | 12 months
  Proportion of subjects achieving greater than 2 point reduction in NASH activity score (NAS) across at least two separate histological components of the NAS score (steatosis, inflammation and ballooning) and no worsening of fibrosis stage.
Biomarker Endpoint | 12 months
  Correlation between presence or absence of histological NASH and combined magnetic resonance (MR) measures and serum cytokeratin 18 (CK18) levels at baseline and 12 month follow-up.

SECONDARY OUTCOMES:
Resolution of NASH: Proportion of subjects achieving "not NASH" histological diagnosis | 12 months
  Proportion of subjects achieving "not NASH" histological diagnosis at the end of the study.
Reduction in mean NAS | 12 months
  decrease in overall histological activity as measured by reduction in mean NAS.
Decrease in steatosis | 12 months
  Decrease in NAS score
Composite decrease in weight | 12 months
  Decrease in BMI, weight and waist circumference.
Composite Quality of Life (QOL) Measures | 12 months
  Change in generic health-related and weight-specific QOL measures Pediatric Quality of Life Inventory and Impact of Weight on Quality of Life (IWQOL-Kids©)).
Liver enzymes | 12 months
  Decrease in serum alanine (ALT) & asparate aminotransferase (AST), gamma-glutamyl trans-peptidase (GGT) level.
Liver enzymes | 12 months
  Normalization of ALT (defined as <26 U/L for males and <22 U/L for females).

CONTACTS AND LOCATIONS:
Overall Officials: Stavra Xanthakos, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States